CLINICAL TRIAL: NCT01523093
Title: An Open Label, Balanced, Randomised, Two-treatment, Two-period, Two-sequence, Single-dose, Crossover Bioavailability Study Comparing Ondansetron 8 mg Orally Disintegrating Tablets of OHM Laboratories Inc (A Subsidiary of Ranbaxy Pharmaceuticals Inc,) With Zofran ODT® 8 mg Orally Disintegrating Tablets (Containing 8 mg of Ondansetron) of GlaxoSmithKline in Healthy, Adult, Human, Male Subjects Under Fasting Condition.
Brief Title: Bioequivalence Study of Ondansetron Orally Disintegrating Tablets 8mg Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Sponsor
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 108_ONDAN_06
Record Dates: First submitted 2012-01-27; First posted 2012-02-01 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
MeSH Terms: interventions — Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zofran ODT (Active Comparator): Zofran ODT (Ondansetron) orally disintegrating tablets 8mg Manufactured By Cardinal Health, Blagrove, Swindon, Wiltshire, UK SN58RU
  Interventions: Drug: Ondansetron
- Ondansetron Orally Disintegrating Tablets (Experimental): Ondansetron 8 mg Orally Disintegrating Tablets Manufactured By OHM Laboratories Inc (A subsidiary of Ranbaxy Pharmaceuticals Inc, USA)
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: Ondansetron — Orally Disintegrating Tablets 8mg

SUMMARY:
The purpose of this study is to compare the single-dose oral bioavailability of Ondansetron 8 mg orally disintegrating tablets of OHM Laboratories Inc (A subsidiary of Ranbaxy Pharmaceuticals Inc, USA) with Zofran ODT® 8 mg orally disintegrating tablets of GlaxoSmithKline, USA in healthy, adult, human, male subjects under fasting condition.

DETAILED DESCRIPTION:
The study was conducted as an open label, balanced, randomised, two-treatment, two-period, two-sequence, single-dose, crossover bioavailability study comparing Ondansetron 8 mg orally disintegrating tablets of OHM Laboratories Inc (A subsidiary of Ranbaxy Pharmaceuticals Inc, USA) with Zofran ODT® orally disintegrating tablets (containing 8 mg of ondansetron) of GlaxoSmithKline in healthy, adult, human, male subjects under fasting condition.

During each period of the study after an overnight fast of at least 10 hours, a single oral dose of either test or reference product was administered by placing the tablet on tongue till it dissolved and then swallowed it using 240 mL of drinking water at ambient temperature under supervision of a medical officer.

During the course of the study, safety parameters including vital signs, clinical examination, medical history and clinical laboratory safety tests (hematology, biochemical, serology parameters and urine analysis) were assessed and laboratory parameters of hematology and biochemistry were repeated at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Were in the age range of 18-45 years.
* Were neither overweight nor underweight for his height as per the Life Insurance Corporation of India height/weight chart for non-medical cases.
* Had voluntarily given written informed consent to participate in this study.
* Were of normal health as determined by medical history and physical examination of the subjects performed within 21 days prior to the commencement of the study.

Exclusion Criteria:

* Had history of allergy or hypersensitivity to ondansetron, related drugs or any other serotonin receptor blocker drugs.
* Had history of dizziness, seizures or extrapyramidal symptoms.
* Had history of urticarial reaction or rash on exposure to any drug.
* Had history of anaphylaxis or angina (chest pain).
* Had history of hepatitis, constipation or phenylketonuria.
* Had history of recurrent episodes of headache.
* Had history of bronchospasm, asthma or shortness of breath.
* Had history of hiccups.
* Had any evidence of organ dysfunction or any clinically significant deviation from the normal, in physical or clinical determinations.
* Had presence of disease markers of HIV 1 or 2, Hepatitis B or C viruses or syphilis infection.
* Had presence of values which were significantly different from normal reference ranges and/or judged clinically significant for haemoglobin, total white blood cells count, differential WBC count or platelet count.
* Was positive for urinary screen testing of drugs of abuse (opiates or cannabinoids)
* Had presence of values which were significantly different from normal reference ranges and/or judged clinically significant for serum creatinine, blood urea nitrogen, serum aspartate aminotransferase (AST), serum alanine aminotransferase (ALT), serum alkaline phosphatase, serum bilirubin, plasma glucose or serum cholesterol.
* Had clinically abnormal chemical and microscopic examination of urine defined as presence of RBC, WBC (> 4/HPF), epithelial cells (> 4/HPF), glucose (positive) or protein (positive).
* Had clinically abnormal ECG or Chest X-ray.
* Had history of serious gastrointestinal, hepatic, renal, cardiovascular, pulmonary, neurological or haematological disease, diabetes or glaucoma.
* Had history of any psychiatric illness, which might have impair the ability to provide written informed consent.
* Was regular smokers who smoked more than 10 cigarettes daily or have difficulty abstaining from smoking for the duration of each study period.
* Had history of drug dependence or had excessive alcohol intake on a habitual basis of more than 2 units of alcoholic beverages per day (1 unit equivalent to half pint of beer or 1 glass of wine or 1 measure of spirit) or had difficulty in abstaining for the duration of each study period.
* Used any enzyme modifying drugs within 30 days prior to Day 1 of this study.
* Had participated in any clinical trial within 12 weeks preceding Day 1 of this study.
* Subjects who, through completion of this study, had donated and/or lost more than 350 mL of blood in the past 3 months.

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2006-07; Primary Completion 2006-07 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) and Peak Plasma Concentration (Cmax) of Ondansetron | 0, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 16, 20 and 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Pharmacology Unit, Majeedia Hospital (2nd Floor), New Delhi, New Delhi, India

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html